CLINICAL TRIAL: NCT00660569
Title: Utilization Patterns of Pulmicort HFA in Real Life Practice
Brief Title: Utilization Patterns of Pulmicort in Real Life Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Mónica Tafalla/Medical Science Director, AstraZeneca
Other Study IDs: NIS-RES-PUL-2007/1
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Asthma
Keywords: asthma treatment; utilization; real life practice
MeSH Terms: conditions — Asthma; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Asthmatic patients with a diagnose of at least 12 months of duration before study inclusion, previously treated with Pulmicort chlorofluorocarbons (CFC) who have changed their treatment to Pulmicort HFA

SUMMARY:
The purpose of this study is to identify the potential issues during short and mid term utilization of Pulmicort hydro fluoroaklane (HFA) pressurized metered-dose inhaler (pMDI)and describe associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic patients with a diagnose of at least 12 months of duration before study inclusion
* Patients previously treated with Pulmicort CFC who have changed their treatment to Pulmicort HFA

Exclusion Criteria:

* Disability that, from investigator point of view, prevent from complying the follow up schedule
* To have participated in any clinical study in the past 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population treated by General Practitioner, Pneumologists or Paediatricians
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2008-01; Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Nuevo Rivero, Study Director — AstraZeneca MC SpainEpidemiologyValue Demonstration Unit
Locations (10):
- Spain (10):
  - Research Site, Barcelona, Barcelona
  - Research Site, Sabadell, Barcelona
  - Research Site, Alcorcón, Madrid
  - Research Site, Leganés, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, San Sebastián de los Reyes, Madrid
  - Research Site, Murcia, Murcia
  - Research Site, Olivares, Sevilla
  - Research Site, Toledo, Toledo
  - Research Site, Fuentes de Ebro, Zaragoza